CLINICAL TRIAL: NCT06134700
Title: Low Pressure Versus Standard Pressure Pneumoperitoneum in Laparoscopic Nephrectomy: A Prospective Randomised Controlled Trial
Brief Title: Low Pressure Versus Standard Pressure Pneumoperitoneum in Laparoscopic Nephrectomy
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Institute of medicine, Maharagjung medical campus (Other)
Responsible Party: Principal Investigator, Anjit Phuyal, Dr, Institute of medicine, Maharagjung medical campus
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Other
Other Study IDs: MaharagjungMC
Record Dates: First submitted 2023-10-14; First posted 2023-11-18 (Actual); Last update posted 2023-11-18 (Actual); Status verified 2023-11

CONDITIONS: Non-Functioning Kidney; Renal Cell Carcinoma
MeSH Terms: conditions — Carcinoma, Renal Cell | interventions — Laparoscopy

STUDY DESIGN:
Who Masked: Participant
Masking Description: Participants will be blinded.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Low pressure pneumoperitoneum laparoscopic nephrectomy (Experimental): Pneumoperitonuem Pressure of 8 - 10 mmHg
  Interventions: Procedure: Laparoscopic Surgery
- Standard pressure pneumoperitoneum laparoscopic nephrectomy (Active Comparator): Pneumoperitonuem Pressure of 12 - 15 mmHg
  Interventions: Procedure: Laparoscopic Surgery

INTERVENTIONS:
Procedure: Laparoscopic Surgery — * Surgery will then proceed at either 8 - 10 or 12 - 15 mmHg pneumoperitoneum pressure depending on study group the patient falls into
  * Port Placement
  * Reflection of colon
  * Isolation of ureterogonadal packet
  * Upper pole dissection
  * Hilar dissection
  * Vessel clipping and division
  * Dissection of kidney
  * Delivery through either Pfannenstiel or iliac fossa incision

SUMMARY:
Laparoscopic nephrectomies are commonly performed these days and are considered gold standard for both benign and malignant diseases as well as for donor nephrectomies. Despite being a widely performed surgery worldwide still there are areas of uncertainties due to lack of evidences. One of such area of dilemma is the optimum pressure of pneumoperitoneum. This study aims to identify if lower pressure of pneumoperitoneum is safe during laparoscopic nephrectomies.

This is a hospital based prospective randomized control study. All the patients undergoing laparoscopic nephrectomies at department of urology and kidney transplant surgery will be eligible for study. Patients will be divided into low pressure or standard pressure pneumoperitoneum by simple random sampling and comparison of various intraoperative and post-operative parameters will be done to assess the safety of low pressure pneumoperitoneum

ELIGIBILITY:
Inclusion Criteria:

* All patients undergoing laparoscopic nephrectomy

Exclusion Criteria:

* Age <18 years
* History of previous abdominal surgeries
* Laparoscopic donor nephrectomies

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 44 (Estimated)
Dates: Start 2023-11-15 (Estimated); Primary Completion 2024-08-15 (Estimated); Study Completion 2024-12-15 (Estimated)

PRIMARY OUTCOMES:
To compare the safety of low pressure versus standard pressure pneumoperitoneum in laparoscopic nephrectomy | 30 days perioperative period
  Complications between two groups will determine the safety of procedure.
To compare the efficacy of low pressure versus standard pressure pneumoperitoneum in laparoscopic nephrectomy | 30 days perioperative period
  Operative time will help to determine efficacy of treatment.

IPD SHARING:
Plan to Share IPD: No